CLINICAL TRIAL: NCT01067144
Title: Stanford Accelerated Recovery Trial (START)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial met futility stopping point
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Assistant Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB-16617; SU-02032010-4882 (Other: Stanford University); VAR0054 (Other: OnCore)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pain; Breast Cancer; Lung Cancer
MeSH Terms: conditions — Pain; Breast Neoplasms; Lung Neoplasms | interventions — Gabapentin; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Control (Placebo Comparator): Active placebo given pre-operatively, followed by inactive placebo for 10 doses post-operatively
  Interventions: Drug: Lorazepam (active control); Drug: Placebo (inactive)
- Gabapentin (Experimental): 1200 mg Gabapentin preoperative dose, 300 mg of Gabapentin 3-times a day postoperative doses for 72-hour post-surgical period.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 1200 mg Gabapentin preoperative dose, 300 mg of Gabapentin 3-times a day postoperative doses for 72-hour post-surgical period.
  Other Names: Fanatrex; Gabarone; Gralise; Neurontin; Nupentin
  Arms: Gabapentin
Drug: Lorazepam (active control) — 0.5 mg Lorazepam (active control) given pre-operatively in a single dose.
  Arms: Control
Drug: Placebo (inactive) — 2 capsules of inactive placebo given 3-times a day post-operatively for the 72-hour post-surgical period.
  Arms: Control

SUMMARY:
The goal of this study is to determine whether administering Gabapentin prior to surgery affects duration of pain and opioid use post-surgery. The investigators aim to compare gabapentin to placebo in a prospective, randomized clinical trial in which patients will be followed post-surgery until pain resolves and opioid use ceases.

DETAILED DESCRIPTION:
Gabapentin was originally developed as an anti-convulsant, but was quickly recognized as a medication with significant analgesic activity in patients with neuropathic pain. More recently it has begun to be appreciated that it may have some benefits in the peri-operative period. Pre-operative Gabapentin reduces preoperative anxiety, early post-operative pain severity, post-operative opioid use and post-operative delirium (presumably through reduced opioid consumption). These same attributes are shared by medications such as NSAIDS and tylenol and the use of peri-operative gabapentin has not permeated the standard of care. Early post-operative pain severity and preoperative anxiety have been implicated in our own research as risk factors for prolonged time to pain resolution and prolonged time to opioid cessation. Since these endpoints are generally synonymous with time to recovery, interventions reducing these times would be seen not just to increase comfort but to actually speed recovery.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 18 to 75
* Undergoing a scheduled surgery
* English speaking
* Ability and willingness to complete questionnaires or use Palm Pilot

EXCLUSION CRITERIA

* Known kidney disease
* Currently receiving gabapentin or (pregabalin) lyrica already
* Cognitive impairment
* Previous history of excessive sedation or adverse reaction to gabapentin (not it was tried but ineffective for nerve pain)
* Coexisting chronic pain > 4/10 disorder in area other than surgical target
* Plan to move out of state
* Condition that would in judgment of team member make patient likely to be lost to follow-up
* Elevated suicidality
* Known pregnancy
* Current symptoms of ataxia, dizziness, or sedation
* Narrow angle glaucoma
* Severe respiratory insufficiency (ie, severe emphysema or chronic obstructive pulmonary disease)
* History of gastric bypass surgery and obstructive sleep apnea requiring continuous positive airway pressure (CPAP)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2010-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Carroll, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Hah J, Mackey SC, Schmidt P, McCue R, Humphreys K, Trafton J, Efron B, Clay D, Sharifzadeh Y, Ruchelli G, Goodman S, Huddleston J, Maloney WJ, Dirbas FM, Shrager J, Costouros JG, Curtin C, Carroll I. Effect of Perioperative Gabapentin on Postoperative Pain Resolution and Opioid Cessation in a Mixed Surgical Cohort: A Randomized Clinical Trial. JAMA Surg. 2018 Apr 1;153(4):303-311. doi: 10.1001/jamasurg.2017.4915. PMID 29238824
- [Derived] Hah JM, Cramer E, Hilmoe H, Schmidt P, McCue R, Trafton J, Clay D, Sharifzadeh Y, Ruchelli G, Goodman S, Huddleston J, Maloney WJ, Dirbas FM, Shrager J, Costouros JG, Curtin C, Mackey SC, Carroll I. Factors Associated With Acute Pain Estimation, Postoperative Pain Resolution, Opioid Cessation, and Recovery: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2019 Mar 1;2(3):e190168. doi: 10.1001/jamanetworkopen.2019.0168. PMID 30821824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1805 patients were assessed for eligibility; 422 were enrolled and randomized.
Groups:
- Control: Active placebo (lorazepam 0.5 mg) given pre-operatively, followed by inactive placebo for 10 doses post-operatively.
Period: Treatment
Arm/Group | Control | Gabapentin
Started | 207 | 215
Completed | 203 | 208
Not Completed | 4 | 7
Not completed — Did not receive allocated intervention | 4 | 7
Period: Follow-up
Arm/Group | Control | Gabapentin
Started | 203 | 208
Intention-to-Treat Analysis Set (Received allocated treatment and had follow-up data.) | 202 | 208
Completed | 144 | 152
Not Completed | 59 | 56
Not completed — Lost to Follow-up | 22 | 12
Not completed — Censored owing to second surgery | 19 | 28
Not completed — Withdrawal by Subject | 18 | 14
Not completed — Surgery cancelled | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Gabapentin | Total
Number analyzed (Participants) | 202 | 208 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.8) | 57.0 (11.7) | 56.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data missing for 1 patient in each group.
  Participants
    number analyzed (Participants) | 201 | 207 | 408
    Female | 123 | 120 | 243
    Male | 78 | 87 | 165

OUTCOME MEASURES:

1. Primary Outcome: Time to Pain Resolution
Description: Time to pain resolution was defined as 5 consecutive reports of "0" average pain at the surgical site (as reported by the patient on a scale of 0-10, with lower scores corresponding to less pain ("0" = no pain) and higher scores corresponding to more pain). Planned call frequency was daily for 3 months, weekly thereafter up to 6 months, and monthly thereafter up to 2 years after surgery.
Time Frame: Up to 2 years
Population: Intention-to-Treat Analysis Set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Gabapentin
Number analyzed (Participants) | 202 | 208
days | 73 [36 to 231] | 84 [36 to 203]

2. Secondary Outcome: Time to Opioid Cessation
Description: Time to opioid cessation was defined as 5 consecutive reports of no opioid use. Planned call frequency was daily for 3 months, weekly thereafter up to 6 months, and monthly thereafter up to 2 years after surgery.
Time Frame: Up to 2 years
Population: Intention-to-Treat Analysis Set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Gabapentin
Number analyzed (Participants) | 202 | 208
days | 32 [9 to 88] | 25 [8 to 53]

3. Secondary Outcome: Count of Participants With Continued Pain at 6 Months
Description: Continued pain was defined as a report of at least "1" average pain at the surgical site (as reported by the patient on a scale of 0-10, with lower scores corresponding to less pain ("0" = no pain) and higher scores corresponding to more pain).
Time Frame: Month 6
Population: Intention-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Gabapentin
Number analyzed (Participants) | 202 | 208
Participants | 37 | 42

4. Secondary Outcome: Count of Participants With Continued Pain at 1 Year
Description: as for outcome 3
Time Frame: Year 1
Population: Intention-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Gabapentin
Number analyzed (Participants) | 202 | 208
Participants | 18 | 21

5. Secondary Outcome: Count of Participants With Continued Opioid Use at 6 Months
Description: Continued opioid use was defined as any report of any continued opioid use at Month 6.
Time Frame: Month 6
Population: Intention-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Gabapentin
Number analyzed (Participants) | 202 | 208
Participants | 4 | 5

6. Secondary Outcome: Count of Participants With Continued Opioid Use at 1 Year
Description: Continued opioid use was defined as any report of any continued opioid use at Year 1.
Time Frame: Year 1
Population: Intention-to-Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Gabapentin
Number analyzed (Participants) | 202 | 208
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Control | Gabapentin
Serious Adverse Events (participants affected / at risk) | 2/202 | 2/208
Other Adverse Events (participants affected / at risk) | 191/202 | 208/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=202) | Gabapentin (N=208)
Postoperative hemodynamic instability (Blood and lymphatic system disorders) | 1 | 0
Hematoma (Blood and lymphatic system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=202) | Gabapentin (N=208)
Leg swelling (General disorders) | 56 | 49
Generalized weakness (General disorders) | 122 | 119
Headache (Nervous system disorders) | 68 | 81
Abdominal pain (Gastrointestinal disorders) | 44 | 30
Diarrhea (Gastrointestinal disorders) | 8 | 11
Dry mouth (Gastrointestinal disorders) | 184 | 192
Constipation (Gastrointestinal disorders) | 147 | 128
Nausea (Gastrointestinal disorders) | 125 | 117
Vomiting (Gastrointestinal disorders) | 55 | 49
Impaired coordination (Nervous system disorders) | 66 | 89
Memory (Nervous system disorders) | 72 | 75
Sore throat (Gastrointestinal disorders) | 113 | 104
Rash (Skin and subcutaneous tissue disorders) | 14 | 27
Visual disturbance (Eye disorders) | 45 | 63
Eye pain (Eye disorders) | 19 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes